CLINICAL TRIAL: NCT01081743
Title: Evaluation de la Mise en Place d'un Auxiliaire d'évaluation Dans la Prise en Charge de la Maladie d'Alzheimer et Des Maladies apparentées en France
Brief Title: Effectiveness of Care Management in Alzheimer Patients
Acronym: AIDALZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Sante Publique, d'Epidemiologie et de Developpement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCB : 2009-A00326-51
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer Disease or Associated Disorder; Mild to Moderately Severe Dementia
Keywords: Alzheimer; Dementia; Mild to moderately severe; New diagnosis; Prevention of behavioural problems
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Social worker (Experimental)
  Interventions: Other: Intervention of the social worker
- Control (No Intervention): Control group is followed-up as usually (usual care)

INTERVENTIONS:
Other: Intervention of the social worker — Systematic home visits and regular follow-ups by phone from a social worker
  Arms: Social worker

SUMMARY:
Context: The French Alzheimer plan 2008-2012 includes the implementation of "disease managers" or social workers, from the onset of the disease, for every patient with a diagnosis of Alzheimer disease or associated disorder. However, previous trials evaluating the efficacy of a systematic intervention for each case from the onset of the disease, including non complex cases, have shown little evidence.

Objective: To evaluate the efficacy of a social worker to prevent behavioural problem for patient with a new diagnosis of Alzheimer disease or associated disorder.

Design and setting: Multicentric cluster randomized control trial. Patients from several memory consultations and specialists (neurologist, psychiatrist or geriatrician) in France are included.

Intervention: In addition to usual care, patients in the intervention group have systematic home visits from a social worker and regular follow-ups by phone over a one-year period. This social worker informs the patient and caregiver, evaluates the needs, gives advices to prevent complications and is a link between the patient and the memory consultation or the specialist. Patient in the control group have absolutely no intervention and are followed-up as usually. In order to not modify the usual care, they have no information on their participation in this trial before the one-year evaluation.

Main outcome measure: NeuroPsychiatric Inventory (NPI) administrated at one year, which evaluates frequency, severity and repercussion of several behavioural problems. Secondary outcomes included disability, cognition, depression, health, quality of life, institutionalization, and resource use.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease or other dementia (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition [DSM IV] criteria of dementia)
* Presence of an informal caregiver
* Mild to moderately severe dementia (MMSE [10-28])
* Diagnosis of dementia made by a specialist ≤ 6 months
* Patient affiliated to the national health insurance system

Exclusion Criteria:

* Institutionalized patient
* Patient on legal guardianship
* Behavioural problem with important clinical repercussion
* Psychotic syndrome
* Severe and unstable general pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-11-24 (Actual); Primary Completion 2013-10-02 (Actual); Study Completion 2013-10-02 (Actual)

PRIMARY OUTCOMES:
NeuroPsychiatric Inventory (NPI) | 1 year
  Evaluation of frequency, severity and repercussion of several behavioural problems

SECONDARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) | 1 year
Apathy Inventory | 1 year
Disablement Assessment for Dementia (DAD) | 1 year
Mini Mental State Examination (MMSE) | 1 year
Global Deterioration Scale (GDS) | 1 year
Montgomery-Asberg Depression Rating Scale (MADRS) | 1 year
Questionnaire Quality of Life - Alzheimer's Disease (QoL-AD) | 1 year
Burden Interview of Zarit | 1 year
Resource utilization in dementia scale (RUD Lite) | 1 year
Medical Outcome Study Short Form 36-item health survey (MOS SF-36) | 1 year
Institutionalization | 1 year
Tiredness scale | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- ISPED (Institut de Santé Publique, d'Epidémiologie et de Développement), Bordeaux, France